CLINICAL TRIAL: NCT04587310
Title: Does Laparoscopic Sleeve Gastrectomy Lead to Barrett's Esophagus, 5-year Esophagogastroduodenoscopy Findings: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Eliana Al Haddad (Other)
Responsible Party: Sponsor-Investigator, Eliana Al Haddad, post-doc research fellow, Jaber Al Ahmad Al Sabah Hospital
Organization: Jaber Al Ahmad Al Sabah Hospital (Other)
Other Study IDs: IJS-S-20-02914
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Laparoscopic Sleeve Gastrectomy — bariatric surgery

SUMMARY:
Introduction Laparoscopic Sleeve Gastrectomy (LSG) is one of the most prevalent approaches to tackle obesity and its co-morbidities. The main complication following the LSG is Gastro-esophageal reflux disease (GERD), with most patients developing worsening symptoms of GERD, and a small number progressing to Barrett's esophagus. This retrospective analysis aims to assess the rate of GERD pre- and post- LSG as well as the rate of progression to Barrett's.

Methods Data was collected from 1639 patients. 92 patients fit our inclusion criteria. Data was then analyzed and summarized against similar literature

ELIGIBILITY:
Inclusion Criteria:

* patients eligible to sleeve gastrectomy that had an EGD pre and 5 years post-op

Exclusion Criteria:

* missing or implausible data, had multiple surgeries, and suffered from the common post-sleeve complications, such as leaks, strictures and hiatal hernias

Ages: 24 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Data was collected from 1639 patients. 92 patients fit our inclusion criteria. Data was then analyzed and summarized against similar literature
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
endoscopy performed on patients | 5 years
  endoscopy will be performed on patients 5 years after undergoing sleeve gastrectomy due to the fact that sleeve tends to lead to reflux which causes dysplasia of esophageal cells, which eventually can lead to barrett's esophagus and cancer.